CLINICAL TRIAL: NCT06202768
Title: Role of the Intrapartum Grobman Nomogram in the Indication of Attempted Vaginal Delivery After Cesarean Section
Acronym: GPP
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, COTTEZ Charlotte, post-resident, Central Hospital, Nancy, France
Other Study IDs: 2023PI211
Record Dates: First submitted 2024-01-01; First posted 2024-01-12 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Vaginal Delivery
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Main population: History of cesarean section Vertex singleton gestation At term (at least 37 weeks of gestation)
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — data collection : age, gestational age, BMI, history of vaginal delivery after cesarean section, indication for cesarean section, preeclampsia for this pregnancy, the cervix dilatation, position in the pelvis, cervix consistency

SUMMARY:
The rate of pregnant patients with a history of cesarean section is increasing. Caesarean section is a surgery which is not without risk and in particular concerning the risk of uterine rupture and malplacentation during a new pregnancy.

Considering the outcome of a new birth following a cesarean section is not easy. There is no reliable score to predict the success rate of vaginal delivery with a history of scarred uterus. The aim of our study would be to validate the intrapartum Grobman nomogram within the population of the Nancy University Hospital and thus to target the population for whom vaginal delivery could be offered.

ELIGIBILITY:
Inclusion Criteria:

* Vertex singleton pregnancy
* Full-term delivery (beyond 37 weeks)
* A history of cesarean section (segmental transverse scar)

Exclusion Criteria:

* Fetal death in utero

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population of women who gave birth at the Nancy maternity ward and met the inclusion criteria, from January 2014 to January 2021.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Modified Grobman score | per-partum, 9 months
  calculate Grobman score according to different criteria. If the score is high, the probability of vaginal delivery is high. This a score which calculates probability of vaginal delivery thanks to 11 parameters (maternal âge, BMI, previous vaginal delivery before and after ceasection, recurring indication, gestational age, hypertensive disease of pregnancy, effacement, dilatation, foetal station, labor induction)

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte COTTEZ, Study Director — Hospital, Nancy, France
Locations (1):
- Maternity, Nancy, France